CLINICAL TRIAL: NCT03865628
Title: Ultrasound Evaluation of Fetal Hemodynamics and Its Variations in Small Fetuses Looking for Prognostic Factors of Perinatal Complications
Brief Title: Ultrasound Evaluation of Fetal Hemodynamics and Perinatal Complications
Acronym: PTI'DOP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Centre Hospitalier Universitaire Dijon (Other); University Hospital, Strasbourg, France (Other); Centre Hospitalier Auxerre (Unknown); Hopital Nord Franche-Comte (Other)
Responsible Party: Sponsor
Other Study IDs: API/2017/89
Record Dates: First submitted 2019-03-04; First posted 2019-03-07 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-02

CONDITIONS: Intrauterine Growth Restriction; Small-for-gestational Age
Keywords: Doppler; Ombilical artery; Middel cerebral artery; Ductus venous; Aortic isthmus; Amniotic fluid; Intrauterine Growth Restriction; Small-for-gestational Age; Prognosis
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In case of fetal weight below the 10th centile for gestational age, it is important to distinguish SGA and IUGR. SGA is defined as a fetal weight below the 10th centile. IUGR correspond to a pathologic reduction of growth velocity and it is a major determinant of perinatal mortality and morbidity. Even if SGA have long time been considered to be constitutionally small without adverse outcomes, recent evidence has demonstrated that a proportion of SGA, with normal UA Doppler, could be associated with neonatal adverse outcomes, probably related to a late-onset IUGR. Therefore, it seems essential to differentiate several categories of fetuses presenting abnormal fetal weight or intrauterine growth: fetuses SGA without any Doppler abnormalities, fetuses affected by early or late-IUGR. In case of late-IUGR, an important part of these fetuses is initially considered as PAG with a normal umbilical Doppler.

In case of fetal weight below the 10th centile for gestational age, longitudinal assessment of the fetal weight and umbilical artery (UA) Doppler is recommended. In case of abnormal UA Doppler, Middle Cerebral Artery (MCA) Doppler is recommended to research a "brain-sparing" effect. If UA and MCA Doppler findings seem to become abnormal in the early stages of IUGR, Ductus Venosus (DV) flow abnormalities have been described as a late marker of fetal decompensation related to an acute myocardial impaired relaxation and acidemia which is a major contributor to adverse perinatal outcome and neurological. The aortic isthmus (AoI) Doppler is an indicator of the progression of fetal hemodynamic deterioration in IUGR and recent data confirm that AoI and DV abnormalities are correlated but AoI Doppler abnormalities would occur earlier than DV Doppler. AoI Doppler could identify abnormalities suggestive of right ventricular dysfunction before DV Doppler and anticipate obstetrical management. In conclusion, Doppler examination could not be reduced to UA Doppler in case of SGA and IUGR and require a global examination including MCA and probably DV and AoI Doppler.

That's why fetal growth assessment should not be limited to fetal biometry and umbilical artery Doppler. Thanks to a systematic protocol for Doppler examination based on UA, MCA, DV and Aortic Isthmus (AoI) Doppler, we hope identify these hemodynamic variations in a large cohort of fetuses <10 to improve prenatal assessment of these foetus to and perinatal outcomes, reducing perinatal morbi-mortality.

DETAILED DESCRIPTION:
All women were followed at one referent matron-fetal medicine unit where they delivered or to which they were referred for abnormalities of the fetal growth. Conforming to national guidelines, referent ultrasound scans and longitudinal assessment of the estimated fetal weight (EFW) were performed depending on the EFW. Each eligible woman was given an information sheet concerning the study protocol.

Fetal biometry and Doppler were performed thanks to a standardised protocol based on international guidelines. In all instances, ultrasound examinations were performed by one experienced and certified operators using an ultrasound machine (GE Voluson E8/E10, GE Medical Systems). EFW was calculated from head and abdominal circumferences and femur length using the formula of Hadlock. The reference growth curves was CFEF growth curves.

Pulsed Doppler measurements were performed automatically, based on at least three consecutive waveforms, with angle of insonation as close to 0° as possible and always below 30°. A high-pass filter of 70 Hz was used to record low-flow velocities and to avoid artifacts. The Umbilical Artery (UA)-PI Doppler were measured at the placental insertion of the funicular cord. The Middle Cerebral Artery (MCA)-PI was obtained in a transverse view of the fetal head, at the level of its origin from the circle of Willis, and the cerebroplacental ratio (CPR) was calculated as the ratio MCA-PI / UA-PI. Aortic Isthmus (AoI)-PI was measured at the level of the three vessels and trachea view, placing the gate just before the convergence of the AoI and the arterial duct. Ductus Venosus (DV)-PI was measured in a mid-sagittal or transverse section of the fetal abdomen, positioning the Doppler gate at its isthmic portion. Participation in the study does not lead to any change in practices or additional data.

In order to ensure the reproducibility of the data and to limit the measurement biases, we will perform a second reading of the Doppler to verify the application of the measurement protocol, especially: acquisition, Doppler spectrum and measurements. A first analysis will focus on the first 10 patients included per center and then, a random analysis on 10 patients every 100 patients included.

Regularly, data monitoring will be made by a scientific technician to reduce missing data.

Anonymous sonographic data were automatically extracted from the electronic patient record (Diamm (MICRO6 SARL) or ViewPoint (General Electric Healthcare France)) and compiled into an electronic case report form with demographic, maternal, obstetrical and neonatal data. Regular extraction will allow to test extraction pipeline and statistical test.

Given a 10% prevalence of SGA, an expected inclusion rate with completed data of 90% and the number of births in the several units, a sample size of 1200 newborns was sufficient to identify 20% of adverse perinatal outcome.

Quantitative variables will be described using the following parameters: mean, standard deviation, median, and minimum and maximum values. Qualitative variables will be described by the frequency and proportion of each class. The qualitative variables will be compared by Chi² test or Fisher exact test. Quantitative variables will be compared by a Student test or a Mann & Whitney test. We will focus on describing the temporal dynamics of the cerebro-aortic relationship.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Estimation of the fetal weight less than estimation the 10th percentile

Exclusion Criteria:

* Refusal of parents
* Fetal and vascular malformations
* Fetal anemia

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population correspond to the patients follow up in one of the materno-fetal medicine unit, multidisciplinary reference unit for the diagnosis, the investigation and management of materno-fetal diseases.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Global perinatal morbidity and mortality | 1 month after birth
  Defined by the occurrence of at least one of the following events (composite outcome of the french national epidemiological study "EPIPAGE"):
  * perinatal death
  * stage 3 or 4 intraventricular haemorrhage
  * cystic periventricular leukomalacia
  * hyperoxic retinopathy treated using laser
  * ulcerative necrotizing enterocolitis
  * bronchopulmonary dysplasia

SECONDARY OUTCOMES:
Specific perinatal morbidity and mortality | 1 month after birth
  Defined by the occurrence of at each events belonging of the composite primary outcome.
Early neonatal morbidity | 1 week after birth
  Defined by the occurrence of at least one of the following events (composite TASK FORCE outcome) :
  * fetal metabolic acidosis with pH <7.00 and base excess> 12 mmol / L
  * early onset of severe or moderate neonatal encephalopathy (after 34 weeks of gestational age)
  * cerebral palsy
  * absence of other causes of encephalopathies (traumatic, bleeding disorders, infections, genetics)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meher S, Hernandez-Andrade E, Basheer SN, Lees C. Impact of cerebral redistribution on neurodevelopmental outcome in small-for-gestational-age or growth-restricted babies: a systematic review. Ultrasound Obstet Gynecol. 2015 Oct;46(4):398-404. doi: 10.1002/uog.14818. PMID 25683973
- [Background] Benavides-Serralde A, Scheier M, Cruz-Martinez R, Crispi F, Figueras F, Gratacos E, Hernandez-Andrade E. Changes in central and peripheral circulation in intrauterine growth-restricted fetuses at different stages of umbilical artery flow deterioration: new fetal cardiac and brain parameters. Gynecol Obstet Invest. 2011;71(4):274-80. doi: 10.1159/000323548. Epub 2011 Feb 24. PMID 21346314
- [Background] Figueras F, Benavides A, Del Rio M, Crispi F, Eixarch E, Martinez JM, Hernandez-Andrade E, Gratacos E. Monitoring of fetuses with intrauterine growth restriction: longitudinal changes in ductus venosus and aortic isthmus flow. Ultrasound Obstet Gynecol. 2009 Jan;33(1):39-43. doi: 10.1002/uog.6278. PMID 19115231
- [Background] Cruz-Martinez R, Figueras F, Hernandez-Andrade E, Oros D, Gratacos E. Changes in myocardial performance index and aortic isthmus and ductus venosus Doppler in term, small-for-gestational age fetuses with normal umbilical artery pulsatility index. Ultrasound Obstet Gynecol. 2011 Oct;38(4):400-5. doi: 10.1002/uog.8976. Epub 2011 Jul 26. PMID 21567514
- [Background] Baschat AA. Planning management and delivery of the growth-restricted fetus. Best Pract Res Clin Obstet Gynaecol. 2018 May;49:53-65. doi: 10.1016/j.bpobgyn.2018.02.009. Epub 2018 Mar 1. PMID 29606482